CLINICAL TRIAL: NCT06994936
Title: An Open-label, Randomized, Parallel-group, Single-dose Relative Bioequivalence Study of Sonelokimab Administered Subcutaneously Either by a Prefilled Syringe or an Autoinjector in Healthy Adults
Brief Title: An Open-label Study in Healthy Adults to Evaluate the Relative Bioequivalence of a Single-dose Administration of Sonelokimab Either by a Prefilled Syringe or an Autoinjector
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MoonLake Immunotherapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: M1095-HV-102
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Relative Bioequivalence
MeSH Terms: interventions — sonelokimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonelokimab via a PFS (Experimental)
  Interventions: Drug: Sonelokimab
- Sonelokimab via an AI (Experimental)
  Interventions: Drug: Sonelokimab

INTERVENTIONS:
Drug: Sonelokimab — sonelokimab 120 mg administered subcutaneously via a PFS
  Arms: Sonelokimab via a PFS
Drug: Sonelokimab — sonelokimab 120 mg administered subcutaneously via an AI
  Arms: Sonelokimab via an AI

SUMMARY:
This is a study to confirm the relative bioequivalence of sonelokimab administered subcutaneously via a prefilled syringe (PFS) or an autoinjector (AI) in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 18 and 55 years of age with suitable veins for cannulation or repeated venipuncture .
* Participants must have a body weight greater than 40 kg and body mass index (BMI) between 21 and 30 kg/m2, inclusive.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physician examination, laboratory tests, and cardiac monitoring.
* Female participants are eligible to participate if they are not pregnant or breastfeeding
* Male participants must be willing to use a condom when sexually active with a partner of childbearing potential during the study, unless surgically sterile.

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
* History of clinically significant infections.
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric.
* History of hypersensitivity, intolerance, or severe adverse reaction to any drug compound, any history of anaphylaxis or angioedema, or any history of severe food allergy/intolerance requiring systemic treatment.
* Participants with transaminase and liver function test results outside of the normal reference range, following a confirmatory test, if appropriate
* Participants with other clinically significant laboratory test results that are likely to introduce additional risk factors or interfere with the study procedures or interpretation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2025-06-05 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Comparison of pharmacokinetics (PK) of an AI versus PFS administered single dose of sonelokimab | 64 days
  To compare the PK of an AI versus PFS administered single-dose of sonelokimab in terms of maximum concentration (Cmax)
Comparison of pharmacokinetics (PK) of an AI versus PFS administered single dose of sonelokimab | 64 days
  To compare the PK of an AI versus PFS administered single-dose of sonelokimab in terms of area under the time concentration curve to infinite time (AUC0-inf)
Comparison of pharmacokinetics (PK) of an AI versus PFS administered single dose of sonelokimab | 64 days
  To compare the PK of an AI versus PFS administered single-dose of sonelokimab in terms of area under the time concentration curve from time zero to timepoint with last measurable concentration (AUC0-t)

SECONDARY OUTCOMES:
Assessment of safety and tolerability | 64 days
  To assess the safety and tolerability of AI and PFS administered sonelokimab by treatment emergent adverse events (TEAEs), serious adverse events (SAEs) and adverse events of special interest (AESIs)
Evaluation of the impact of injection site location on PK | 64 days
  Evaluation of the impact of injection site location on PK by capturing the relative bioavailability (F%) for thigh injection of sonelokimab compared to abdomen
Evaluation of the impact of injection site location on PK | 64 days
  Evaluation of the impact of injection site location on PK by capturing the relative bioavailability (F%) for upper-arm injection of sonelokimab compared to abdomen
Evaluation of the impact of injection site location on PK | 64 days
  Evaluation of the impact of injection site location on PK by capturing the relative bioavailability (F%) for thigh injection of sonelokimab compared to upper arm
Immunogenicity of sonelokimab | 64 days
  Description of the prevalence of antidrug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site, London, United Kingdom